CLINICAL TRIAL: NCT06531070
Title: Effects of Different Nitrate Formulations on Strength and Endurance Performance in Recreationally Trained Adults
Brief Title: Nitrate Formulations and Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Greenwich (Other)
Collaborators: Crown Sport Nutrition (Industry)
Responsible Party: Principal Investigator, Fernando Naclerio, Professor, University of Greenwich
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: NITR 24.10.23; CEAR ILD (Other: university of Greemwoch)
Record Dates: First submitted 2024-07-23; First posted 2024-07-31 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-07

CONDITIONS: Nitrate; Nitrate/Citrulline; Placebo
MeSH Terms: interventions — Nitrates; Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nitrate (Experimental): A gel providing 600 mg (9.6 mmol) of nitrate.
  Interventions: Dietary Supplement: Nitrate
- Nitrated and citrulline (Experimental): A gel, providing 600mg of nitrate (9.6 mmol) and 6 g of citrulline-malate
  Interventions: Dietary Supplement: Nitrate
- Placebo (Placebo Comparator): Placebo in gel format providing negligible amount of nitrate
  Interventions: Dietary Supplement: Nitrate

INTERVENTIONS:
Dietary Supplement: Nitrate — A four-day supplementation period, separated by one week including a 3-day washout period between conditions will be applied before conducting strength and endurance assessments
  Days 1 to 3 the randomly assigned supplement (N, NC, or PLA) will be ingested 2 hr before a standard low-volume training session including 3 sets of 8 to 10 reps of squat and deadlift using a very light load (e.g., own body mass) and flexibility exercises following by 5 min of running at self-paced intensity rated as light (12) with the rating of perceived exertion Borg Scale.
  Day 4: the assigned supplement will be ingested 2.5 h before the assessments
  Assessment of strength and endurance will be conducted
  Other Names: Nitrated and citrulline; Placebo

SUMMARY:
this study compares the acute effects of Nitrate and Nitrate plus citrulline supplementation on physical performance in recreationally trained males and females. This is a cross-over within-participant comparison design concluding three arms (i) 600 mg of Nitrate (N), ii) 600 mg Nitrate and Citrulline (NC) and (iii) Placebo (PL).

Conditions N, NC and PL will be tested one week apart, considering a minimum washout period of 72 hours.

Dependent variables:

* Number of completed repetitions to failure in squat using 75% of 1RM.
* Ventilatory thresholds (VT1) and (VT2) and Vo2 max from a progressive to exhaustion running test (PGT)
* Lactate post (within 1 min of having completed the PGT)
* Rating of perceived exertion (RPE) by the Borg 6-to-20-point scale recorded every 2 min and at the end of the PGT.
* Heart rate associated with VT1, VT2, and Vo2max - Heart rate maximum.
* Maximal aerobic speed (MAS): calculated from the average speed of the last 2 minutes of the PGT.
* time limit test at MAS (conducted after 15 min of having completed the PGT)

DETAILED DESCRIPTION:
Aim:

To analyse and compare the acute effect of two different nitrate formulations on strength and endurance performance in young recreationally trained individuals. In a cross-over within-participant comparison design the participants will be assigned either to ingest (i) 600 mg of Nitrate (N), ii) 600 mg Nitrate and Citrulline (NC) and (iii) Placebo (PL).

Design: Cross-over randomised controlled within participant design including one group undertaking three different treatment conditions.

1. Nitrate (N) providing 600 mg (9.6 mmol) of Nitrate (NO-3).
2. Nitrate + Citrulline (NC) providing 600 mg (9.6 mmol) of Nitrate (NO-3) and 6 g of citrulline-malate.
3. Placebo (PLA) Participants (15 or higher) Inclusion criteria: (a) males and females 18-40 years of age; (b) physically active participants with experience in resistance training performing squat and endurance running as habitual exercises (c) free from musculoskeletal limitations or injuries, (d) agree not to ingest any other supplement during the study.

Exclusion criteria: (a) a history of various metabolic conditions or diseases; (b) use of a variety of medications, including but not limited to those with androgenic and/or anabolic effects and/or nutritional supplements known to affect training outcomes such as creatine, proteins, etc. within 6 weeks before the beginning of the study, (c) current use of tobacco products.

All participants must provide written informed consent by the Declaration of Helsinki. The University ethics committee must approve procedures before starting with the data collection.

Procedures Day 0: Familiarization with the testing procedures including the progressive test to determine the 1RM value in Squat.

Diet Record: Each participant will complete a 1-week diet record using a food frequency questionnaire (FFQ). This questionnaire consists of questions relating to the weekly consumption of different types of food, to estimate energy consumption and the nutritional composition of the reported diets. Participants were instructed to maintain their habitual diet throughout the study. If any change in diet patterns is identified, the participants were dropped from the study.

Supplementation protocol:

Days 1 to 3 Supplements (N, NC, or PLA) will be ingested 2 hr before a standard low-volume training session including 3 sets of 8 to 10 reps of squat and deadlift using a very light load (e.g., own body mass), and flexibility exercises following by 5 min of running at self-paced intensity rated as light (RPE 12). This routine can be completed at home.

Day 4: supplements will be ingested 2.5 hours before the assessments.

The three conditions Nitrate (N) Nitrate + Citrulline (NC) and Placebo (PL) will be tested one week apart, considering a minimum washout period of 72 hours, a strategy that has previously been used in studies with a similar design.

All participants will be following an identical training week in each of the three treatment conditions.

Dependent variables:

o Number of completed repetitions in a singular set to failure in a squat with 75% of 1RM.

Lactate Post (within 1 min of having completed the squat) 15 min rest Progressive to exhaustion on a treadmill (PGT)

* Ventilatory thresholds (VT1) and (VT2)
* Vo2 max
* Lactate post (within 1 min of having completed the PGT)
* Rating of perceived exertion (RPE) using the Borg 6-to-20-point scale recorded every 2 min and at the end of the PGT.
* Heart rate associated with VT1, VT2, and Vo2max - Heart rate maximum.
* Maximal aerobic speed (MAS): calculated from the average speed of the last 2 minutes of the PGT.

  15 min rest
* Maximal Aerobic Speed test (no cortex).
* Lactate pre (15 min post PGT)
* The participants should run until exhaustion at the previously determined MAS (e.g. 19.8 km/h)
* RPE after 1 minute and at the end
* Heart rate every 1 minute and at the end
* Lactate post (within 1 minute of having completed the test

ELIGIBILITY:
Inclusion Criteria

* Physically active participants with experience in resistance training performing squats and endurance running as habitual exercises
* Free from musculoskeletal limitations or injuries
* Agree not to ingest any other supplement during the study.

Exclusion Criteria

* History of various metabolic conditions or diseases
* Use of a variety of medications, including but not limited to those with androgenic or anabolic effects or nutritional supplements known to affect training outcomes such as creatine, proteins, etc. within 6 weeks before the beginning of the study
* Current use of tobacco products.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Strength | Day 4, 2.5 hours after ingesting the supplement
  Ten maximum repetitions set in back squat using 75% of the previously determined maximal strength determined by the maximum amount of kg lifter in one sigulare repetitions
Maximum oxygen consumption (Vo2max) | through study completion up to 3 weeks
  The highest level of oxygen determined during a progressive to exhaustion running test on a treadmill (PGT)

SECONDARY OUTCOMES:
Ventilatory thresholds (VT1) and (VT2) | 15 minutes after completing the strength test
  ventilatory thresholds using a gas analyser during a progressive to exhaustion running test on a treadmill (PGT)
lactate | through study completion up to 3 weeks
  lactate concentration
Heart Rate | through study completion up to 3 weeks
  Heart Rate response to endurance PGT test
Rate of Perceived Exertion | through study completion up to 3 weeks
  Perception of effort

OTHER OUTCOMES:
Maximal Aerobic Speed | through study completion up to 3 weeks
  the speed at which the Vo2 maximum is determined during the PGT test

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Naclerio, Principal Investigator — University of Greenwich
Locations (1):
- Sparrows Farm, Eltham, London, United Kingdom